CLINICAL TRIAL: NCT02550301
Title: Prospective Pilot Study- Does Mean Platelet Volume Change With Clopidogrel in Patients With Stable Angina Undergoing Percutaneous Coronary Intervention?
Brief Title: Does Mean Platelet Volume Change With Clopidogrel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-8707
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Stable Angina
Keywords: mean platelet volume
MeSH Terms: conditions — Angina, Stable | interventions — Mean Platelet Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood in EDTA collection tubes to measure Mean Platelet Volume
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mean Platelet Volume: 4 blood samples (1 pre procedure before clopidogrel loading) and 3 after Percutaneous Coronary Intervention will be drawn to assess the MPV
  Interventions: Other: Mean Platelet Volume

INTERVENTIONS:
Other: Mean Platelet Volume — Ten milliliters (mls) of blood will be drawn from eligible, consented patients at the time of the admission, collected in ethylenediamine tetraacetic acid (EDTA) tubes, and tested for CBC. Platelets have an average life span that can vary from 8-10 days or 10-36 days. To minimize this bias, three additional MPV samples will be collected on day 1, day 7 and day 30 post PCI.

SUMMARY:
Platelets play a major role in thrombus formation and platelet size, measured by Mean Platelet Volume (MPV) correlates with platelet activity. MPV is increased in patients with Myocardial Infarction (MI) and is an independent predictor of adverse events in patients with ST Elevation Myocardial Infarction (STEMI) . Data on MPV in patients with stable angina is limited.

Aspirin and clopidogrel are antiplatelet agents administered routinely to patients undergoing PCI and are required for stent patency. MPV is not known to be affected by low dose Aspirin. Treatment with clopidogrel is thought to reduce MPV in-vitro but the magnitude of this reduction in MPV is unclear, especially in patients with stable angina undergoing PCI. An inverse correlation also exists between MPV and platelet count .

The investigators aim to assess if a change occurs in MPV (∆ MPV) after routine clopidogrel administration in patients with stable angina undergoing PCI.

DETAILED DESCRIPTION:
This is a prospective, observational study. The investigators aim to conduct this pilot study to assess if there is a change in MPV (∆ MPV) after routine clopidogrel in patients with stable angina undergoing PCI.

Reduced responsiveness to clopidogrel (otherwise known as clopidogrel resistance) is well documented. Clopidogrel resistance can result in adverse long term effects including stent thrombosis and mortality. Diagnosis of clopidogrel resistance requires special analyzers and reagents . There are potential cost factors involved with the analyzers and reagents used for testing resistance. There are no known clinical or biochemical markers of clopidogrel resistance.

If our pilot study results demonstrate that MPV does change (∆MPV) after clopidogrel, then a prospective trial can be conducted in future to correlate ∆MPV with clopidogrel resistance measured by analyzer tests. This could establish ∆MPV as a potential cheap, effective biochemical marker for clopidogrel resistance.

If the investigators are successful in demonstrating a change in MPV with clopidogrel, our pilot study will facilitate conducting future larger studies to demonstrate correlation between ∆MPV and clopidogrel resistance. This could establish ∆MPV as a potential cheap, effective biochemical marker for clopidogrel resistance with resultant benefit to subjects and the institution.

All clopidogrel naive patients with stable angina symptoms who are electively listed for coronary angiography and PCI at Peter Munk Cardiac Centre (PMCC), Toronto General Hospital (TGH), will be included in this pilot study. This pilot study will be conducted in compliance with the protocol, Good Clinical Practice (GCP) and University Health Network (UHN) policy

Study hypothesis. The investigators hypothesize that MPV values remain the same after clopidogrel in patients with stable angina undergoing PCI and aim to disprove the hypothesis

Study Design This prospective pilot study will include consecutive clopidogrel naïve patients with stable angina symptoms, who are electively listed for coronary angiography and PCI at Peter Munk Cardiac Centre (PMCC), Toronto General Hospital (TGH), will be prospectively included in this pilot study. These patients are given a routine loading dose of clopidogrel 600milligrams (mg) followed by a daily dose of clopidogrel 75mg daily after they undergo PCI (as per protocol for all patients who undergo PCI). Complete Blood Count (CBC) is performed routinely in patients prior to the loading dose of clopidogrel (day 0) and on one occasion post PCI as per UHN standard of care. MPV and platelet count are automatically generated during analysis of CBC.

Ten milliliters (mls) of blood will be drawn from eligible, consented patients at the time of the admission, collected in ethylenediamine tetraacetic acid (EDTA) tubes, and tested for CBC. Platelets have an average life span that can vary from 8-10 days or 10-36 days12. To minimize this bias, three additional MPV samples will be collected on day 1, day 7 and day 30 post PCI.

The samples will be analyzed within 2 hours of venipuncture to minimize artefactual increase in MPV with prolonged exposure to EDTA in the collection tubes .

Change in MPV (∆MPV) and change in platelet count (∆Platelet count) will be calculated as follows:

* MPV = MPV on admission - Mean MPV after clopidogrel
* Platelet count = Platelet count on admission - Mean Platelet count after clopidogrel These results will be correlated with adverse events (readmission and MI) at 30 days by collecting data regarding readmission and cardiac blood tests (for MI) from the electronic patient record (EPR) system online. The universal definition of MI will be adhered to .

Platelet inhibition occurs within 2 hours of a loading dose but reaches a steady state from 3 to 7 days. Repeated samples will ensure the effect of a steady level of clopidogrel on MPV and reduce bias.No change in intervention or medication will occur-all patients will receive treatment according to the UHN standard of care. No randomization or blinding is involved in this pilot study.

The expected duration of participation will be up to 1 month after the index procedure as repeat blood tests are required at day 7 and day 30 after the procedure and adverse events are assessed at day 30.

Patients discharged on the day of the procedure need to return for blood tests the following day, on day 7 and day 30 after the PCI (3 visits). Patients discharged on the day after the procedure will need to return for blood tests on day 7 and day 30 after the PCI (2 visits).

This will involve travel time (approximately 1 hour each way) and time to give the blood sample (30 minutes inclusive of waiting time) equal to a total of 2.5 hours for each visit. Patients will have an overall time commitment of 7.5 hours for 3 visits or 5 hours for 2 visits.

Statistics MPV is automatically analyzed (on a CBC sample) by the Abbott CELL-DYN Sapphire@ analyzer at the TGH laboratory.

The sample size was estimated using the formula:

Z = 1.96 for 95% Confidence Interval (CI) σ = standard deviation (SD) of the outcome variable = 0.219 fl for MPV (Hematology Laboratory Quality Control (QC) for MPV analyzed by Abbott CELL-DYN Sapphire@ (8.46 fl). E (5%) = desired margin of error

In order to ensure that the 95% confidence interval estimate of the MPV in adults with stable angina undergoing PCI is within 0.219 femtolitre (fl) of the true mean MPV, a sample size of 74 patients is required for this pilot project.

Assuming an attrition rate of 30%, a sample size of 100 patients would be required. The formula has taken into account the QC mean obtained for the Abbott CELL-DYN Sapphire@. An attrition rate of 30% was taken into account for patients who may not be able to return for the repeat blood tests.

In addition to determining if MPV changes after clopidogrel or not, ∆MPV will be correlated with the presence of clopidogrel using Receiver Operating Curves (ROC) as will ∆Platelet count. The study will be terminated on completion of collection of 4 blood samples at pre-specified time points in 74 patients (actual calculated sample size) with stable angina undergoing angiography and PCI.

All eligible patients (as per the inclusion criteria) will be included in the trial.

Only persons involved in this pilot study (i.e. PI, Co-PI, research fellows and research nurse) will have access to the source data and documents which will be maintained in a secure location at the PMCC site. Any electronic data will be on specific UHN designated on-site computers, password protected and only accessible to the designated research team.

Review and Assessment of adverse events Adverse effects are not expected at the time of blood collection. A designated contact telephone number for the research nurse will be made available to the participating patients in the event of rare adverse effects such as fainting at the time of blood collection, bruising or infection at the access site.

Consent process Patients will be consented prior to the procedure - the background of the proposed study and the relative benefits and risks of the study will be clearly explained to the patient prior to the procedure on the day. If the patient's native language is not English or the patient does not speak/understand English, then a UHN designated native language translator will be involved for purposes of consent. Patients must sign the consent form prior to enrollment. A UHN prototype consent form prototype will be used for this purpose.

Co-ordinated Approval Process for Clinical Research (CAPCR) form has been submitted for and approved by the Research Ethics Board (REB)

Financing: Funding will be obtained (internally) from the Cardiology Division, PMCC, TGH.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Able to attend for follow up blood tests
* Able to provide written informed consent

Exclusion Criteria:

* <18 years of age
* Unable to attend for follow up blood tests on days 1, 7 and 30
* Already on clopidogrel at least 1 day prior to presenting for angiography/PCI
* Those who undergo only diagnostic angiography
* History of Myocardial Infarction (MI) in last 1 year
* Anemia (Hb<100)
* Abnormal (low or high out of range) platelet counts
* Diabetes Mellitus
* Known liver disease
* Known severe renal impairment (eGFR <30ml/min/1.73m2)
* Known pregnancy
* On Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) or steroids
* Known connective tissue disease
* Acute ongoing infections or bleeding
* On oral anticoagulant treatment in the last 1 week
* Pro-coagulant blood disorder
* Known immunosuppressed states
* Treatment with GpIIb/IIIa inhibitor in the last week prior to presentation
* Patients involved in other trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who are clopidogrel naïve, electively listed for coronary angiography and Percutaneous Intervention (PCI) at PMCC, Toronto General Hospital (TGH), will be prospectively enrolled in this pilot study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in MPV (∆MPV) with clopidogrel in stable angina patients undergoing PCI. | 30 days

SECONDARY OUTCOMES:
Change in Platelet count (∆ platelet count) with clopidogrel in stable angina patients | 30 days
Correlation between ∆MPV and adverse events (readmission and Myocardial Infarction) at 30 days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD,FRCPC, Principal Investigator — University Health Network, Toronto

REFERENCES:
- [Background] Martin JF, Shaw T, Heggie J, Penington DG. Measurement of the density of human platelets and its relationship to volume. Br J Haematol. 1983 Jul;54(3):337-52. doi: 10.1111/j.1365-2141.1983.tb02109.x. PMID 6860588
- [Background] Pizzulli L, Yang A, Martin JF, Luderitz B. Changes in platelet size and count in unstable angina compared to stable angina or non-cardiac chest pain. Eur Heart J. 1998 Jan;19(1):80-4. doi: 10.1053/euhj.1997.0747. PMID 9503179
- [Background] Huczek Z, Kochman J, Filipiak KJ, Horszczaruk GJ, Grabowski M, Piatkowski R, Wilczynska J, Zielinski A, Meier B, Opolski G. Mean platelet volume on admission predicts impaired reperfusion and long-term mortality in acute myocardial infarction treated with primary percutaneous coronary intervention. J Am Coll Cardiol. 2005 Jul 19;46(2):284-90. doi: 10.1016/j.jacc.2005.03.065. PMID 16022956
- [Background] Jagroop IA, Mikhailidis DP. Mean platelet volume is an independent risk factor for myocardial infarction but not for coronary artery disease. Br J Haematol. 2003 Jan;120(1):169-70. doi: 10.1046/j.1365-2141.2003.03983_4.x. No abstract available. PMID 12492596
- [Background] Shah B, Valdes V, Nardi MA, Hu L, Schrem E, Berger JS. Mean platelet volume reproducibility and association with platelet activity and anti-platelet therapy. Platelets. 2014;25(3):188-92. doi: 10.3109/09537104.2013.793794. Epub 2013 Jun 20. PMID 23786366
- [Background] Goncalves SC, Labinaz M, Le May M, Glover C, Froeschl M, Marquis JF, O'Brien E, Shukla D, Ruchin P, Sookur D, Ha A, So D. Usefulness of mean platelet volume as a biomarker for long-term outcomes after percutaneous coronary intervention. Am J Cardiol. 2011 Jan 15;107(2):204-9. doi: 10.1016/j.amjcard.2010.08.068. Epub 2010 Dec 2. PMID 21129717
- [Background] Gasparyan AY, Ayvazyan L, Mikhailidis DP, Kitas GD. Mean platelet volume: a link between thrombosis and inflammation? Curr Pharm Des. 2011;17(1):47-58. doi: 10.2174/138161211795049804. PMID 21247392
- [Background] Bessman JD, Williams LJ, Gilmer PR Jr. Mean platelet volume. The inverse relation of platelet size and count in normal subjects, and an artifact of other particles. Am J Clin Pathol. 1981 Sep;76(3):289-93. doi: 10.1093/ajcp/76.3.289. PMID 7282629
- [Background] Snoep JD, Hovens MM, Eikenboom JC, van der Bom JG, Jukema JW, Huisman MV. Clopidogrel nonresponsiveness in patients undergoing percutaneous coronary intervention with stenting: a systematic review and meta-analysis. Am Heart J. 2007 Aug;154(2):221-31. doi: 10.1016/j.ahj.2007.04.014. PMID 17643570
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Matetzky S, Shenkman B, Guetta V, Shechter M, Beinart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Circulation. 2004 Jun 29;109(25):3171-5. doi: 10.1161/01.CIR.0000130846.46168.03. Epub 2004 Jun 7. PMID 15184279
- [Background] Bautista AP, Buckler PW, Towler HM, Dawson AA, Bennett B. Measurement of platelet life-span in normal subjects and patients with myeloproliferative disease with indium oxine labelled platelets. Br J Haematol. 1984 Dec;58(4):679-87. doi: 10.1111/j.1365-2141.1984.tb06115.x. PMID 6240280
- [Background] Endler G, Klimesch A, Sunder-Plassmann H, Schillinger M, Exner M, Mannhalter C, Jordanova N, Christ G, Thalhammer R, Huber K, Sunder-Plassmann R. Mean platelet volume is an independent risk factor for myocardial infarction but not for coronary artery disease. Br J Haematol. 2002 May;117(2):399-404. doi: 10.1046/j.1365-2141.2002.03441.x. PMID 11972524
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432